CLINICAL TRIAL: NCT03476174
Title: MMP-01: Pilot Study Evaluating Activity of the Combination of Anti-PD-1 Antibody With High Dose IL-2 in Metastatic Melanoma
Brief Title: Anti-PD-1 Antibody With HD IL-2 in Metastatic Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Accrual
Sponsor: Ralph Hauke (Other)
Collaborators: Nebraska Cancer Specialists Methodist Estabrook Cancer Center (Other); Prometheus Laboratories (Industry)
Responsible Party: Sponsor-Investigator, Ralph Hauke, Chief of Hematology and Oncology, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN-MMP-MEL16-261
Record Dates: First submitted 2018-03-16; First posted 2018-03-23 (Actual); Results first posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab and HD Interleukin 2 (Experimental): Pembrolizumab 200 mg IV over 30 minutes; Day 1 of each cycle 3 weeks (21 days) for 2 cycles. IL-2 600,000 IU/kg2 IV over 15 minutes every 8 hours for up to 14 doses over 5 days; Days 1-5 = Cycle 1; 9 days of rest in between; Days 15-19 = Cycle 2
  Interventions: Drug: Pembrolizumab; Drug: Interleukin-2

INTERVENTIONS:
Drug: Pembrolizumab — Subjects will receive 200 mg pembrolizumab every 3 weeks for two cycles. Cycle length is 21 days (i.e., 3 weeks). On the last day of Cycle 2 (+/- 3 days), disease status will be assessed via imaging.
  Other Names: Keytruda
Drug: Interleukin-2 — Following the pembrolizumab treatment, HD IL-2 treatment will commence. After completing the 2 cycles of pembrolizumab, High Dose Interleukin-2 (HD IL-2) will be administered. This will require a hospital stay of at least 5 days for each treatment cycle. Established guidelines will be followed for safely administering HD-IL-2 and managing toxicities from this treatment. Two treatment cycles will be administered, Cycle 2 being separated from Cycle 1 by approximately 9 days after completion (assuming subject has recovered from Cycle 1 adequately to proceed with Cycle 2). Four weeks after completion of the 2 cycles (called a course of HD IL-2 therapy), disease status will be monitored via CT of the chest and abdomen/pelvis using revised RECIST guidelines
  Other Names: High Dose IL-2

SUMMARY:
The primary objective of this single arm phase 2 trial is to assess the response rate [complete response (CR) + partial response (PR)] of sequential therapy of pembrolizumab followed by HD IL-2 in subjects with stage IV malignant melanoma. Response assessment will be performed after pembrolizumab therapy, and response reassessment will be performed after HD IL-2 therapy using revised RECIST 1.1.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status of 0-1 within 28 days prior to registration (Appendix 1).
* Life expectancy of 6 months or greater as determined by the site investigator.
* Histologically-confirmed diagnosis of unresectable stage IV or metastatic melanoma not amenable to local therapy.
* Measurable disease, defined as at least 1 tumor that fulfills the criteria for a target lesion according to RECIST 1.1 (Section 9), and obtained by imaging within 28 days prior to registration for protocol therapy.
* < 2 lines of prior therapy for metastatic melanoma. Cannot have received prior therapy with HD IL-2. May have had one prior line of therapy that included a check point inhibitor.
* Prior systemic cancer treatment must be completed at least 21 days prior to first dose of study drug and the subject must have recovered from all reversible acute toxic effects of the regimen (other than alopecia or vitiligo) to Grade ≤ 1 or baseline.
* Not received radiation therapy within 21 days of initiation of study treatment, and the measurable disease must have been outside of the radiation port.
* Demonstrate adequate organ function. All screening labs to be obtained within 28 days prior to registration.

  * WBC ≥ 3,000/L
  * ANC ≥ 1,000/L
  * Hgb ≥ 9g/dL
  * Plt ≥ 100 × 10(9)/L
  * Serum creatinine ≤ 1.5 mg/dL
  * Calculated creatinine clearance ≥ 40 mL/min; if serum creatinine > 1.5 mg/dL
  * Total Bilirubin ≤ 1.5 × upper limit of normal (ULN)
  * Direct Bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 x ULN
  * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT)≤ 2.5 × ULN or ≤ 5 x ULN for subjects with known hepatic metastasis
  * International Normalized Ratio (INR) ≤ 1.5 × ULN; For subjects receiving warfarin or LMWH, the subjects must, in the site investigator's opinion, be clinically stable with no evidence of active bleeding while receiving anticoagulant therapy. The INR for these subjects may exceed 1.5 × ULN if that is the goal of anticoagulant therapy.
* Adequate baseline pulmonary function test (PFT) (FEV1 > 2 L or ≥ 75% of predicted for height and age).
* Documented left ventricular ejection fraction (LVEF) of > 45%, testing is required in patients with:

  * Age ≥ 60 years old
  * Clinically significant atrial and or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block
  * History of coronary revascularization or ischemic symptoms
* Archival tissue (from the primary tumor or metastases) is mandatory if available for correlative studies. If archived tumor tissue is not available, the patient does not need to undergo a biopsy to obtain tissue and is still eligible for study.
* Females of childbearing potential must have a negative serum pregnancy test within 3 days prior to registration. NOTE: Females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months
* Females of childbearing potential and males must be willing to abstain from heterosexual activity or to use 2 forms of effective methods of contraception from the time of informed consent until 120 days after treatment discontinuation. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method.
* Male subjects who are not surgically sterile (vasectomy) must agree to use an adequate method of contraception. Male subjects with female sexual partners who are pregnant, possibly pregnant or who could become pregnant during the study must agree to use condoms from the first dose of study drug through 120 days after the last dose of study therapy. Total abstinence for the same study period is an acceptable alternative.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Active infection requiring systemic therapy
* Pregnant or breastfeeding. NOTE: breast milk cannot be stored for future use while the mother is being treated on study.
* Known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer, or other cancer for which the subject has been disease-free for at least five years.
* Active central nervous system (CNS) metastases. NOTE: if prior metastasis but treated and clinically stable for 1 month after treatment are eligible. Subjects with 3 or fewer brain metastases that are less than 1 cm in diameter and asymptomatic are eligible.
* Surgery within 4 weeks prior to study treatment except for minor procedures. NOTE: Hepatic biliary stent placement is allowed.
* Uncontrolled or poorly-controlled hypertension (> 160 mmHg systolic or > 100 mmHg diastolic for > 4 weeks) despite standard medical management.
* Serious or non-healing wound, ulcer, or bone fracture within 28 days prior to initiation of study treatment.
* Any Grade 3-4 GI bleeding within 3 months prior to initiation of study treatment.
* History of deep vein thrombosis, pulmonary embolism, or any other significant thromboembolism (venous port or catheter thrombosis or superficial venous thrombosis are not considered "significant") during the 3 months prior to initiation of study treatment.
* Any arterial thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within 6 months prior to initiation of study treatment.
* Gross hemoptysis within 2 months of initiation of study treatment.
* Has any condition that, in the opinion of the investigator, might jeopardize the safety of the patient or interfere with protocol compliance.
* Has any mental or medical condition that prevents the patient from giving informed consent or participating in the trial.
* Known hypersensitivity to pembrolizumab or IL-2 or any of their components.
* Known history of active tuberculosis.
* Concurrent systemic steroid therapy with doses above physiologic level.
* History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with anti-phospholipid syndrome, granulomatosis with polyangiitis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.

  * Subjects with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible for this study.
  * Subjects with controlled Type I diabetes mellitus on a stable dose of insulin regimen may be eligible for this study.
  * Subjects with a history of celiac disease may be eligible if controlled with diet.
* Treatment with any investigational agent within 21 days prior to initiation of study treatment and the subject must have recovered from the acute toxic effects of the regimen.
* Prior organ transplant including allogeneic transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Hauke, MD, Principal Investigator — Nebraska Cancer Specialists Methodist Estabrook Cancer Center
Locations (1):
- Nebraska Cancer Specialists, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab and HD Interleukin 2
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: One subject was registered to this study before termination by the funder
Arm/Group | Pembrolizumab and HD Interleukin 2
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 53 [53 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) from 0-5 that describes a patient's level of functioning where 0=Fully active, able to carry on all pre-disease performance without restriction and 5=Dead
  Participants
    ECOG PS =0 | 1
    ECOG PS =1 | 0

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Assess the response rate [complete response (CR) + partial response (PR)] of sequential therapy of pembrolizumab followed by HD IL-2 in subjects with stage IV malignant melanoma. Response assessment will be performed using revised RECIST 1.1
Time Frame: 12 months
Population: Due to the early termination of the study by the funder, data for this objective was not formally analyzed. Individual subject responses are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab and HD Interleukin 2
Number analyzed (Participants) | 1
Participants
  Complete Response | 1
  Partial Response | 0
  Stable Disease | 0
  Progressive Disease | 0

2. Secondary Outcome: Assess Adverse Events
Description: Assess adverse events via CTCAE v4.03
Time Frame: 12 months
Measure: Number; unit: participants experiencing adverse event
Arm/Group | Pembrolizumab and HD Interleukin 2
Number analyzed (Participants) | 1
participants experiencing adverse event
  ENCEPHALOPATHY GR 4 | 1
  HEPATIC FAILURE GR 4 | 1
  HYPOXIA GR 4 | 1
  RESPIRATORY FAILURE GR 4 | 1
  CREATININE INCREASED GR 3 | 1
  HYPOTENSION GR 3 | 1
  ALLERGIC REACTION GR 2 | 1
  DIARRHEA GR 2 | 1
  DIZZINESS GR 2 | 1
  HOARSENESS GR 2 | 1
  TREMOR GR 2 | 1
  WEIGHT LOSS GR 2 | 1
  EDEMA LIMBS GR 1 | 1
  EDEMA TRUNK GR 1 | 1
  LETHARGY GR 1 | 1
  WEIGHT GAIN GR 1 | 1

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Measure Progression-Free Survival (PFS) using revised RECIST guideline (version 1.1) after completion of 2 cycles of pembrolizumab and 2 cycles of HD IL-2 in all the subjects enrolled in the study. PFS is defined as the time from treatment initiation until objective tumor progression or death.
Time Frame: 12 months
Population: Due to the early termination of the study by the funder, data for this objective was not collected or analyzed
Arm/Group | Pembrolizumab and HD Interleukin 2
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival (OS)
Description: Measure overall survival (OS) at 12 months in subjects with stage IV malignant melanoma who showed a response [stable disease (SD), complete response (CR) or partial response (PR)] following completion of 2 cycles of pembrolizumab and 2 cycles of HD IL-2. OS is defined as time from treatment initiation until death from any cause
Time Frame: 12 months
Population: Due to the early termination of the study by the funder, data for this objective was not collected or analyzed
Arm/Group | Pembrolizumab and HD Interleukin 2
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From screening until subject discontinuation due to termination of the study at nine months.
Arm/Group | Pembrolizumab and HD Interleukin 2
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab and HD Interleukin 2 (N=1)
ENCEPHALOPATHY GR 4 (Nervous system disorders) | 1 (1)
HEPATIC FAILURE GR 4 (Hepatobiliary disorders) | 1 (1)
HYPOXIA GR 4 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY FAILURE GR 4 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab and HD Interleukin 2 (N=1)
CREATININE INCREASED GR 3 (Investigations) | 1 (1)
HYPOTENSION GR 3 (Cardiac disorders) | 1 (1)
ALLERGIC REACTION GR 2 (Immune system disorders) | 1 (1)
DIARRHEA GR 2 (Gastrointestinal disorders) | 1 (1)
DIZZINESS GR 2 (Nervous system disorders) | 1 (1)
HOARSENESS GR 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
TREMOR GR 2 (Nervous system disorders) | 1 (1)
WEIGHT LOSS GR 2 (Investigations) | 1 (1)
EDEMA LIMBS GR 1 (General disorders) | 1 (1)
EDEMA TRUNK GR 1 (General disorders) | 1 (1)
LETHARGY GR 1 (Nervous system disorders) | 1 (1)
WEIGHT GAIN GR 1 (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early by the funder after a single subject accrual and no formal analysis was conducted for any study endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/74/NCT03476174/Prot_SAP_000.pdf